CLINICAL TRIAL: NCT07214246
Title: Investigating the Role of Follicular Fluid microRNAs in Ovarian Aging and Assisted Reproductive Success
Brief Title: Follicular Fluid microRNAs in Ovarian Aging and Reproduction
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: The IVF Center at Winter Park (Unknown)
Responsible Party: Sponsor
Other Study IDs: STUDY00008057
Record Dates: First submitted 2025-10-08; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Aging; In Vitro Fertilisation (IVF) Treatment; InVitro Fertilization; In Vitro Fertilization Outcome
Keywords: IVF; In vitro fertilization; Follicular fluid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Interventions — No interventions for participants

SUMMARY:
The purpose of this study is to investigate the role of exosomal microRNAs (miRNAs) in follicular fluid (FF) as biomarkers of ovarian aging and predictors of in vitro fertilization (IVF) outcomes. The goal is to identify noninvasive molecular markers that correlate with oocyte quality and reproductive potential, particularly in women of advanced maternal age.

DETAILED DESCRIPTION:
There is a substantial gap in understanding how these miRNAs operate in humans, especially in a non-invasive or minimally invasive context.

Specifically:

* The role of exosomal miRNAs in follicular fluid (FF) in human ovarian aging is not well defined.
* Few studies have directly compared miRNA expression profiles in FF across age groups using high-throughput sequencing.
* There is limited evidence linking specific FF miRNAs to oocyte quality or IVF success rates.
* No validated non-invasive biomarkers based on FF exosomal miRNA currently exist for predicting IVF outcomes, especially in women of advanced reproductive age.

This study seeks to address these knowledge gaps by identifying and validating exosomal miRNA signatures in FF that are associated with maternal age and IVF outcomes. The most relevant preliminary data come from preclinical rodent studies performed by our research team:

* miRNA profiling in aged vs. young mouse ovarian tissues demonstrated clear age-associated changes in miRNA expression.
* Gene target analyses revealed that these miRNAs are likely to regulate critical signaling pathways involved in ovarian aging (e.g., FoxO, mTOR, PI3k/Akt).
* These results support the biological plausibility that similar miRNA changes could occur in human follicular environments and impact oocyte competence.

Although direct human data from FF is not yet available, the team has validated methods for exosome isolation from biofluids, miRNA sequencing, and in vitro assays. These tools are now being applied to the human FF samples collected during IVF cycles, making this study a logical and feasible extension of our previous work.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF treatment due to male factor infertility or nonovarian causes.
* Age groups: younger women <31 years and older women >38 years.
* Regular menstrual cycles.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Minors (under 18 years) and women aged 32-37 years
* Diagnosis of polycystic ovarian syndrome (PCOS).
* History of recurrent pregnancy loss.
* Presence of endometriosis.
* Diagnosis of ovarian insufficiency.
* Metabolic disorders (e.g., diabetes).
* History of ovarian surgery or chemotherapy.
* Any condition that might impact follicular fluid quality or IVF outcomes.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing IVF treatments.
Study Population: Potential participants will be screened and identified during their initial consultation and scheduling for IVF treatment at The IVF Center. Medical records and patient history will be reviewed to screen for eligibility based on inclusion and exclusion criteria. Women who meet all inclusion criteria and none of the exclusion criteria will be invited to participate and consented for the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Identify exosomal miRNAs using RNA sequencing | 1 year
  Identify differentially expressed exosomal miRNAs in the follicular fluid of younger (<31 years) versus older (>38 years) women undergoing IVF using small RNA sequencing.
Validate and assess miRNA for IVF | 1 year
  Validate the expression of selected miRNAs in an independent sample set and assess their correlation with clinical IVF parameters, including oocyte maturity, fertilization, and embryo development.
Determine molecular pathways regulated by age | 1 year
  Use bioinformatic analysis and in vitro functional assays to determine the molecular pathways regulated by age associated miRNAs, particularly those involved in follicular development, hormone signaling, and cellular aging.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Masternak, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States